CLINICAL TRIAL: NCT04578054
Title: Benefit of the FLYing Transport of Patients Requiring Mobile Intensive Care Unit
Acronym: FLY-MICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR CNRS 6024 LaPSCo, Clermont-Ferrand, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020 BOUILLON MINOIS Fly Micu
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Stress, Psychological; Emergency Medicine, Transport; Critical Care
Keywords: Stress, Psychological; emergency Medicine, transport; critical care
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Flying transport — Patient care who requires flying transport

SUMMARY:
Patient care who requires fast and intensive care by a mobile intensive care unit in a rescue helicopter is a common practice in Auvergne since more than 3 years. Indeed, a complete team (nurse and emergency physician) is on Dragon 63 and HeliSMUR 63 (SMUR = emergency medical services ). There are multiple fields of action, with a primary rescue activity (patient care directly at the site of the operation) but also secondary transport (transfer of patients from one hospital to another). This allows a reduction in transport time and therefore unavailability of the MICU team in general hospitals, which are in short supply of attending physicians. In addition, this allows patients to be repatriated to the Clermont-Ferrand University Hospital Center, which is the reference center for many pathologies and has the Level 3 adult and pediatric Trauma Center.

DETAILED DESCRIPTION:
This is an observational study using a REDCap® questionnaire via an internet link, which will be distributed by any means (institution mailing lists via a referent, flash codes distributed to physicians, etc.).

The questionnaire will assess the type of medicalisation, the type of activity, the different hours of intervention, the age, the type and the severity of the patient's disease, the type of care practiced and the stress of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Every Emergency Physician that participate to the Helicopter rescue

Exclusion Criteria:

* Every Emergency Physician non-voluntary to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Physician
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Stress | Day 1
  stress level will be assessed by Visual Analog Scale (VAS) from 0 to 10 (0 the lowest stress and 10 the highest)

SECONDARY OUTCOMES:
Severity of the disease | Day 1
  Severity of the disease that need MICU team for the care measure by Classification Clinique des Malades aux Urgence CCMU scale (1 to 5 ; 1 is the lowest problem and 5 the severest ; + P : Psychiatric + D : death at the arrival, no reanimation)
Duration of the care | Day 1
  Every schedules of the care : departure from Clermont-Ferrand University Hospital, arrival at the victim, departure from the accident or take care place, arrival at Clermont-Ferrand university hospital, time of the patient transmission, time of disponibility

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France